CLINICAL TRIAL: NCT05276024
Title: Evaluation of the IFuse Bedrock Technique in Association with Posterior Lumbosacral Fusion with Iliac Fixation.
Status: Recruiting | Type: Observational
Sponsor: Polyclinique Bordeaux Nord Aquitaine (Other)
Collaborators: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-ORT03
Record Dates: First submitted 2022-02-21; First posted 2022-03-11 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Sacroiliitis; Sacroiliac; Fusion; Lumbosacral; Fusion; Spine Deformity
Keywords: Sacroiliac joint pain; Sacroiliac joint fusion; Bedrock technique; Open posterior lumbosacral fusion; Spine deformties
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- iFuse Bedrock technique: Multilevel lumbar fusion procedure with additional sacroiliac joint stabilization using the iFuse-3D system
  Interventions: Device: iFuse Bedrock technique

INTERVENTIONS:
Device: iFuse Bedrock technique — Lumbosacral arthrodesis on 2 or more spinal segments (including at least L4, L5 and S1 vertebrae) associated with a sacroiliac fusion procedure according to the Bedrock technique using the iFuse 3D system and iliac fixation.

SUMMARY:
The purpose of this study is to describe the impact of the iFuse Bedrock technique to decrease post-operative pains in patients who underwent multilevel posterior lumbosacral fusion.

DETAILED DESCRIPTION:
This study is a multicentric, post-marked clinical investigation to assess the efficacy of the iFuse Bedrock technique to avoid post-operative pains in patients who underwent open posterior multilevel lumbosacral fusion. Subjects will be monitored for lumbar pains (Oswestry score, VAS, SF-12 questionnaire) and sacroiliac joint pains (provocative tests) up to 12 months after initial procedure. A single CT-scan acquisition will be performed at 12 months to detect any iFuse system-related abnormality (implants loosening or breakages).

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled for open posterior lumbosacral arthrodesis (including at least the following three vertebrae: L4, L5 and S1) associated with a sacroiliac fusion procedure and iliac fixation (thoracolumbar fusion procedures extended to sacrum are eligible in the study);
* Insertion of at least 1 iFuse-3D implant according to the iFuse Bedrock technique (uni- and bilateral insertion are eligible);
* Subject who preoperatively responded positively to pain provocation tests for SIJ dysfunction with or without a positive SIJ infiltration test;
* Patient with a degenerative sacroiliac joint disease requested a fusion procedure;

Exclusion Criteria:

* Major osteoporosis (DEXA scan > 3);
* Any previous history of sacroiliac joint fusion or any surgical procedure involving a S2-iliac fusion;
* Subjects requested a SIJ fusion without the iFuse-3D device or iFuse-3D not inserted according to the manufacturer instruction (Bedrock technique);
* Subjects with a medical or surgical contraindication preventing the intervention from being performed or potentially interfering in the interpretation of the data collected (neurologic condition, local or systemic infection, any known allergy to surgical implants, psychiatric diseases, ...);
* Currently pregnant or planning pregnancy;
* Prisoner or a ward of the state;
* Subject no willing to participate in the study;
* Subject not affiliated to a social security insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants enrolled in the study are adult subjects who underwent an open posterior lumbosacral fusion procedure with additional sacroiliac joint fusion according to the iFuse Bedrock technique (insertion of the iFUSE-3D implant). Lumbosacral fusion involved at least the following vertebrae : L4, L5 and S1.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in self-reported Oswestry Disability Index (ODI) at 12 months | 12 months
  A decrease of 16 points in the ODI score at 12 months compared to the preoperative score is expected in order to demonstrate a 30% effecacy of the iFuse Bedrock technique in reducing postoperative pain.

SECONDARY OUTCOMES:
Change from baseline in sacroiliac joint pain provocation tests. | During 12 months
  The number of positive SIJ pain provocation tests (Östgaard test, Faber test, Gaenslen test, Lasegue test, Compression, Long ligament test) performed at 3, 6 and 12 months will be compared against baseline (preoperative).
Assessment of the Oswestry Disability Index | 3 and 6 months
  Change from baseline in self reported Oswestry Disability Index (ODI) score at 3 and 6 months.
Improvement of back and leg pains at 3, 6 and 12 months compared to preoperative scores | 3, 6 and 12 months
  Back and leg pain intensity self-report will be assessed before and after initial procedure for each patient (at 3, 6 and 12 months) using a 0 to 10 visual analog scale (0: no pain ; 10: most imaginable pain).
Change in Patient's quality of life | 3, 6 and 12 months
  Change from baseline in self reported 12-Item Short Form Survey (SF-12) score at 3, 6 and 12 months.
Proportion of subjects with postoperative SIJ fusion failure | 12 months
  Proportion of subjects with SIJ fusion failure on CT scan as interpreted by the investigator
Impact of iFuse Bedrock technique on Pelvic Incidence | During 12 months
  Measurement of postoperative Pelvic Incidence (PI) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Pelvic Incidence is the angle between the line perpendicular to the S1 endplate from the midpoint of the endplate and the connecting line from the midpoint of the S1 endplate to center of the femoral head.
Impact of iFuse Bedrock technique on Pelvic Tilt | During 12 months
  Measurement of postoperative Pelvic Tilt (PT) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Pelvic Tilt is the angle between the connecting line from the midpoint of the S1 endplate to the center of the femoral head and the vertical line.
Impact of iFuse Bedrock technique on Sacral Slope | During 12 months
  Measurement of postoperative Sacral Slope (SS) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Sacral Slope is the angle between the tangent and the horizontal line of S1 endplate.
Impact of iFuse Bedrock technique on Lumbar Lordosis | During 12 months
  Measurement of postoperative Lumbar Lordosis (LL) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Lumbar Lordosis is the angle between the L1 upper endplate and the S1 upper endplate.
Impact of iFuse Bedrock technique on Thoracic Kyphosis | During 12 months
  Measurement of postoperative Thoracic Kyphosis (TK) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Thoracic Kyphosis is the angle between the T4 upper endplate and the T12 lower endplate.
Impact of iFuse Bedrock technique on the Odontoid Hip Axis | During 12 months
  Measurement of postoperative Odontoid Hip Axis (OD-HA) using EOS stereography at 3, 6 and 12 months compared to baseline.
  Odontoid Hip Axis is the angle between the vertical and the highest point of the odontoid process (dens) connecting to the centre of the acetabulum (bi-coxo-femoral axis)
Impact of iFuse Bedrock technique on the T1 pelvic angle | During 12 months
  Measurement of postoperative T1 pelvic angle (TPA) using EOS stereography at 3, 6 and 12 months compared to baseline.
  TPA is the angle between the line from centroid of T1 to the femoral head axis and the line from femoral head axis to middle of the S1 endplate
Proportion of subjects with iFuse-3D implant-related complications | 12 months
  Proportion of subjects with any of the following complications related to the iFuse-3D implant : malposition of the implant (intra-operative evaluation), loosening, displacement, abnormal bone reaction, breakage or any other complication directly related to the insertion or use of the iFuse-3D implant.
Incidence of any serious adverse events | During 12 months
  Record of any intra and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jean Charles Le Huec, M.D., PhD, Principal Investigator — VERTEBRA Institute, Polyclinique Bordeaux Nord Aquitaine
Locations (2):
- France (2):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpitaux Universitaires de Marseille, Marseille

IPD SHARING:
Plan to Share IPD: No